CLINICAL TRIAL: NCT00918320
Title: Phase 2 Single- Arm Studies of Temozolomide in Combination With Topotecan in Refractory and Relapsed Neuroblastoma and Other Paediatric Solid Tumours
Brief Title: Studies of Temozolomide in Combination With Topotecan in Refractory and Relapsed Paediatric Solid Tumours
Acronym: TOTEM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: St. Anna Kinderkrebsforschung (Other); Catholic University of the Sacred Heart (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSET 2008/1378
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Neuroblastoma; Brain Tumors; Solid Tumors
Keywords: Temozolomide; Topotecan; paediatric solid tumours; Miscellaneous other solid tumours
MeSH Terms: conditions — Neuroblastoma; Brain Neoplasms | interventions — Temozolomide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Toptecan + temozolomide (Experimental)
  Interventions: Drug: Temozolomide/Hycamtin (Topotecan)

INTERVENTIONS:
Drug: Temozolomide/Hycamtin (Topotecan) — Temozolomide: bottles containing 5 capsules of 5, 20, 100 and 250 mg
  Hycamtin (Topotecan): a lyophilisate for infusion in vials containing 4 mg
  Patients receive during 5 days (Day 1 to Day 5):
  Temozolomide 150 mg/m2/day per os, dose will be adjusted to the closest 5 mg, followed one hour later by Hycamtin(Topotecan) 0.75 mg/m2/day as an intravenous infusion over 30 minutes
  Other Names: Hycamtin:Topotecan

SUMMARY:
The purpose of the study is to determine whether the combination of Hycamtin (Topotecan) and Temozolomide is effective in the treatment of relapsed and refractory neuroblastoma and other paediatric solid tumors.

DETAILED DESCRIPTION:
Current treatments for malignant paediatric solid tumors involve a combination of chemotherapy, surgery and, in certain cases, radiotherapy. This multidisciplinary approach leads to an overall cure of approximately 70%. Nevertheless, cancer mortality remains the leading cause of disease-related death in children and adolescents between 1 and 19 years. This is due to diseases with a poor prognosis, such as metastatic neuroblastoma, sarcoma in soft tissue and bone and brain tumors. New effective treatments must be found in order to continue to increase the cure rate of children and adolescents treated for cancer, as well as to improve the cured patients' quality of life

Neuroblastoma (NB) is a malignant paediatric tumour derived from primordial neural crest cells. This tumor accounts for 8% to 10% of all cancers with a median age of onset of 22 months. The primary tumor may be located in different anatomic sites such as abdomen (65%), thorax (19%), pelvis (2%), and cervix (1%). The strongest prognostic factors are age and stage. Localized NB and those occuring in infants have a 90% survival rate when the biological profile is favorable. Conversely, in case of Myc-N amplification, survival is around 30% after conventional treatment and 70% after intensification. More than 50% of patients have a disseminated tumor at diagnosis, and Stage 4 neuroblastoma in patients older than 1 year of age represents the most frequent form. Neuroblastoma is a chemosensitive tumor. Chemotherapy is indicated in large primary tumours to reduce the volume and attempt a safe surgical resection and to eradicate tumour metastases in disseminated NB. The most frequently used drugs are alkylating and platinum agents (cyclophosphamide, melphalan, cisplatin, carboplatin), topoisomerase II inhibitors (doxorubicin, etoposide) and vinca-alkaloids (vincristine). High-dose chemotherapy (busulfan, melphalan, carboplatin, etoposide) with autologous bone marrow stem cell support is used as a consolidation treatment in patients with metastatic disease, as well as maintenance therapy with retinoid acid. Although such an intensive strategy, the probability of survival of patients over 1 year of age with Stage 4 neuroblastoma is less than 40%. New drugs are urgently needed for patients with recurrent neuroblastoma.

Central nervous system (CNS) tumors as an entity represent the second most frequent malignancy in childhood and adolescents. The incidence rate of childhood primary benign and malignant brain tumors is 3.9 cases per 100,000 person-years, and appears to be increasing. Two thirds of the new cases are in children less than 15 years of age. The morbidity associated with CNS tumors exceeds those of other malignancies and is undoubtedly a result of the neurological and cognitive deficits associated with both the tumor itself and aggressive multimodal therapy. Current treatment involves surgical resection, mostly combined with irradiation and/or chemotherapy. This multidisciplinary approach leads to a cure in about 55% of all brain tumour patients. However, the outcome in small children and certain malignancies, such as high grade astrocytomas, brain stem glioma and atypical teratoid/rhabdoid tumors and metastatic primary neuroectodermal tumors (PNET)/medulloblastoma is still dismal. In addition, treatment with irradiation and/or the combination of different chemotherapeutic agents is at the limit of tolerance inducing renal, hepatic, auditory, or hematological toxicity. Moreover, irradiation to the cerebral hemispheres, especially in small children, induces devastating sequelae. Clinical resistance to anticancer agents is the primary reason for treatment failure in childhood cancer and the development of new agents with a new profile of anti-tumour activity and toxicity is highly warranted.

Other relapsed/refractory non-CNS solid tumors include nephroblastoma, osteosarcoma, Ewing's sarcoma, rhabdomyosarcoma and soft-tissue sarcomas, and rarer tumours, such as hepatoblastoma, retinoblastoma, nasopharyngeal carcinoma, and germ-cell tumours. For most of these tumors, treatment protocols are available for first-line therapy; to a lesser extent, treatment recommendations are proposed in case of relapse. Depending on the disease, type, and localization of relapse, treatment may include combinations of salvage chemotherapy, including high-dose chemotherapy with stem cell rescue, radiotherapy, and surgery.

In several of these diseases, temozolomide (as well as topoisomerase I inhibitors, such as irinotecan and Topotecan) have shown single agent activity and may be used in combination schedules.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed neuroblastoma, brain tumor or other solid tumor (at diagnosis)
* Relapsed or refractory tumors in which correct standard treatment approaches have failed
* No more than 2 lines of prior chemotherapy
* Measurable primary and/or metastatic disease on CT/MRI at least one bi-dimensionally measurable lesion.

For patients with neuroblastoma, measurable disease will be defined by the modified International Neuroblastoma Staging System (Brodeur et al.1993) completed with MIBG scoring.

* Age at inclusion: 6 months to ≤ 20 years
* Lansky play score ≥ 70% or ECOG performance status ≤ 1
* Life expectancy ≥ 3 months
* Adequate organ function:

Adequate haematological function: haemoglobin ≥ 80 g/l, neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 100 x 109/L; in case of bone marrow disease: neutrophils ≥ 0.5 x 109/l and platelets ≥ 75 x 109/l;

Adequate renal function: normal creatinine related to patient's age:

* 0 - 1 year: ≤ 40 µmol/L
* 1 - 15 years: ≤ 65 µmol/L
* 15 - 20 years: ≤ 110 µmol/L Adequate hepatic function: bilirubin ≤ 1.5 x ULN; AST and ALT ≤ 2.5 x ULN (AST, ALT ≤5xULN in case of liver metastases)

  * Wash-out of 4 weeks in case of prior chemotherapy, 6 weeks if treatment included nitrosoureas, 2 weeks in case of vincristine alone; 6 weeks in case of prior radiotherapy (except palliative radiotherapy on non measurable lesions). Patients must have recovered from the acute toxic effects of all prior therapy before enrolment into the study.
  * Patients previously treated with only one of the 2 drugs are eligible.
  * Able to comply with scheduled follow-up and with management of toxicity.
  * All patients with reproductive potential must practice an effective method of birth control while on study. Female patients aged > 12 years must have a negative pregnancy test within 7 days before study treatment.
  * Written informed consent from patient, parents or legal guardian.

Exclusion Criteria:

* Concurrent administration of any other anti-tumour therapy.
* Serious concomitant systemic disorder (for example, active infection including HIV or cardiac disease) that in the opinion of the investigator, would compromise the patient's ability to complete the study.
* History of allergic reaction to the compounds or their solvents.
* History of allergic reaction to Dacarbazine (DITC).
* Galactosemia, Glucose-galactose malabsorption or lactase deficiency.
* Pregnant or breast feeding young women.
* Presence of symptomatic brain metastases in patients with solid non-CNS tumors.

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2009-06; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Response rate | after 2 cycles=8 weeks of therapy

SECONDARY OUTCOMES:
safety and adverse event profile of the combination safety and adverse event | 28 days
time-to-event endpoints: duration of response, time to progressive disease, time to treatment failure and overall survival | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Geoerger, MD, PHD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France